CLINICAL TRIAL: NCT03618563
Title: Developing and Evaluating a Meta-cognitive Intervention Amongst Adolescents With Neuro-development Disabilities
Acronym: FITTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Rosenblum (Other)
Responsible Party: Sponsor-Investigator, Sara Rosenblum, Professor in the Department of Occupational Therapy, Faculty of Social Welfare, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FITTED
Record Dates: First submitted 2018-07-10; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Adolescent Behavior
Keywords: daily function; executive functions
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled and crossover trial to evaluate the efficacy of the treatment among adolescents with EF deficits in their daily performance. The first Intervention Group (A) received the FITTED intervention. After a crossover switching trial, the second Intervention Group (B) received the FITTED intervention in order (Fig 1). An OT performed all four evaluations (Phases 1, 1a, 2, and 3) in similar environmental conditions. Another OT performed the intervention process according to the protocol. The Ethics Committee of the University of Haifa approved the study.
Who Masked: Participant
Masking Description: After the baseline evaluation, participants were randomly assigned to Intervention Group A or B by block randomization. For example, the first participant was allocated to Group A, the second to Group B, third to Group A, and so forth (Jadad 1998). Participants did not know to which group they belonged and had not contact with other participants during all study phases. Further, the OT who performed the participant evaluations was blinded to their treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: functional individualized therapy for teenagers with executive deficits — Intervention to improve self-perceived performance and performance satisfaction in daily activity goals that adolescent selected,

SUMMARY:
Adolescents with neuro-developmental disabilities such as attention deficit hyperactive disorder (ADHD), specific learning disabilities (LD) and developmental coordination disorder (DCD) display functional difficulties in all performance areas (daily functions, learning, playing, leisure activities, and social participation). These problems hinder their ability to perform and participate effectively in everyday life.

Difficulties in meta-cognitive components, particularly Executive Functions (EF), are the underlying mechanisms of these disorders and challenge the functioning of this population. Therefore it is important to refer them to occupational therapists specializing in daily functions and individualized intervention. The proposed model for assessment and therapy, Functional Individualized Therapy for Teenagers with Executive Deficits (FITTED) takes into account the environmental requirements, the person (the adolescent and his pertinent issues), this in accordance with the classifications of the International Classification of Functioning, Disability and Health for Children and Youth (ICF-CY) (WHO, 2007) World Health Organization, the occupational model and dynamic meta-cognitive models. FITTED serves as a basis for an individual evaluation and intervention program that emphasizes the individual's personal strengths and weaknesses in daily functions: Body functions (meta-cognitive - EF and awareness); Activity in various fields and Participation in daily functions. The model will serve as a guide for an intervention program that will be based upon determining functional goals and achievement of these goals through meta-cognitive strategies that will allow adolescents optimal participation in their environments.

DETAILED DESCRIPTION:
Research Aims

1. To construct a theoretical model from existing literature for researchers and clinicians in the field of adolescents with neuro-developmental disorders.
2. To examine the effectiveness of the model through an intervention process that includes assessment and treatment of adolescents with neuro-developmental disorders.

Hypotheses:

The study involved two main groups:

1. The Research Group - a group of adolescents with neurodevelopmental deficiencies (n = 41) divided into two sub-groups: A. Research group A (n = 21) - received treatment immediately after the first assessment. B. Research group B (n = 20) - was reassessed eight weeks after the first assessment (the length of the treatment process), and then received treatment. Both research groups were reassessed at the end of the treatment (second assessment for Group A and third assessment for group B). An additional assessment was performed three months after the end of treatment.
2. The Control Group - typical adolescents (n = 40). Assessed once.

The hypotheses are presented in three stages:

Stage 1:

1. A comparison of the characteristics of the subjects of the research groups (A and B) as a preliminary stage to their unification as one control group (n=41). Hypothesis 1: Differences will not be found in the demographic variables and daily functions when assessed using CHECK the questionnaire and the level of control in EF in the assessment using the BRIEF questionnaire.
2. To examine the change in research group B (n = 20) prior to treatment; Hypothesis 2: Differences will not be found between assessment 1 and assessment 1a before the treatment in the following variables: 2. a. The level of awareness of the subject in execution of daily activities (writing task of copying a passage from the Israeli handwriting quality diagnosis for junior high schools and preparation of a cake and drink from the CCT assessment tool). 2. b. The control of EF (BRIEF questionnaires and a WebNeuro assessment). 2. c. Execution of activities that reflect daily functions (copying a passage from the Israeli handwriting quality diagnosis for junior high schools and preparation of a cake and drink from the CCT diagnostic tool). 2. d. Participation in activities in the home environment, in school and the community (PEM-CY questionnaire).

Stage 2:

Characteristics of the Participants:

1. A comparison of the demographic, personal, family, developmental and educational characteristics of members of the research group (n = 41) with those of the control group (n = 40) and a comparison of the characteristics of the research variables before treatment: Hypothesis 3: Significant differences will be found between the research group and the control group in the demographic personal, family, developmental and educational variables. Hypothesis 4: Significant differences between the research group and the control group, with advantages to the control group in: 4. a. Awareness levels of the adolescent before the execution of daily activities (writing task of copying a passage from the Israeli handwriting quality diagnosis for junior high schools and preparation of a cake and drink from the CCT diagnostic tool). 4. b. Control of EF (BRIEF questionnaires and a WebNeuro assessment). 4. c. Execution of activities that reflect daily functions (copying a passage from the Israeli handwriting quality diagnosis for junior high schools and preparation of a cake and drink from the CCT diagnostic tool). 4. d. Participation in leisure activities and activities in the home environment, in school and the community (PEM-CY questionnaire).
2. Description of treatment goals selected by the participants of the research groups ((n = 41) in the treatment process.

Stage 3:

Effectiveness of the Treatment

1. Examination of the effectiveness of the treatment process within in the research group (n = 41). Hypothesis 5: Significant differences will be found in the research group (n = 41) before and after treatment in : 5. a: The adolescent's level of awareness before performing daily life activities (copying a passage from the Israeli handwriting quality diagnosis for junior high schools and preparation of a cake and drink from the CCT diagnostic tool). 5. b. Control of EF (BRIEF questionnaires and a WebNeuro assessment). 5. c. Performing activities that reflect daily functioning (copying a passage from the Israeli handwriting quality diagnosis for junior high schools and preparation of a cake and drink from the CCT diagnostic tool). 5. d. Participation in activities in the home environment, in school and the community (PEM-CY questionnaire).
2. Examination of the effectiveness of the treatment three months after its completion (n = 41). Hypothesis 6: Differences will be found in the research group before and after treatment, and after a follow-up assessment three months later. 6. a. Control of EF (BRIEF questionnaires). 6. b. Participation in activities in the home environment, in school and the community (through PEM-CY questionnaire).
3. An evaluation of the effectiveness of the treatment in the context of the goals chosen by the adolescent before beginning the treatment:

Hypothesis 7:

7. Differences will be found in the research group in the adolescent's evaluation of his execution in treatment goals as rated with the COPM and GAS before, during and after the treatment, and in the follow-up three months later. (4) A prediction of characteristics of the adolescent's performance after treatment, using meta-cognitive variables that were examined before treatment, as reported by adolescents and parents: Hypothesis 8: The level of control of EF (BRIEF questionnaire and a WebNeuro assessment), and awareness (predictive awareness and awareness to assessment of time) as reported and executed by the adolescent at the beginning of treatment will predict:

8. a. The execution of daily activities such as preparing a cake and a drink as part of the CCT diagnosis. 8. b. The execution of daily activities as assessed through the writing task of copying a passage from the Israeli handwriting quality diagnosis for junior high schools (total time, amount of time the pen was on the paper and in the air). Hypothesis 9: The level of control in EF, as reported by parents at the beginning of treatment through the BRIEF questionnaire, would predict: 9. a. Execution of daily activities such as preparing a cake and a drink as part of the CCT diagnosis - after treatment. 9. b. Execution of daily activities assessed through the writing task of copying a passage from the Israeli handwriting quality diagnosis for junior high schools (total time, amount of time the pen was on the paper and in the air) - after treatment.

Method Participants: Eighty-one adolescents aged 10-18 were accepted to the study according to the inclusion criteria. The participants were divided into two main research groups: the research group (n=41) and the control group (n=40), matched by age and gender. The research group was tested with a Randomized Control Trial (RCT). The participants were found through extensive publication regarding the research. The study included adolescents with deficits in everyday activities according to their parents' reports in the Child Evaluation Checklist (CHECK) questionnaires and EF deficits as reported by their parents in the Behavior Rating Inventory of Executive Function (BRIEF) (score of 65 and higher). Tools: an evaluation was performed to examine the effectiveness of the intervention on daily functions: a Toglia questionnaire (2011) measured awareness; a WebNeuro was used for the neuropsychological testing; and BRIEF questionnaires for parents and the adolescents were used to examine the manifestation of executive functions in daily life. Performance of everyday tasks was measured through a writing task of copying an excerpt from the Israeli handwriting diagnostics for junior high schools, and preparation of a cake and a drink as part of the Children's Cooking Task (CCT).

Participation in the home, at school and in the community were assessed with the Participation Measure and Environment for Children and Youth (PEM-CY) questionnaire. Moreover, the Canadian Occupational Performance Measure - COPM and - Goal Attainment Scaling - GAS were used to assess implementation of the selected treatment goals and satisfaction with performance.. Extensive information on the medical, developmental, personal and educational history and of the subjects was also gathered. Procedure: The study was carried out between the years 2012 and 2015 by two researchers: one performed the assessments, and the chief researcher executed the intervention processes. One group (n=21) was the first to receive the intervention immediately after the primary evaluation, and the second group (n=20) waited during the assessment period, and after a second assessment began treatment. The participants were reassessed after treatment and once again three months later. Data processing: A MANOVA was performed with SPSS-21 to examine the differences between the indices of the research and control groups after their first assessments. Repeated Measures tests were performed in order to measure test hypotheses about differences in the functioning of members of the research group before and after intervention and in the follow-up. Regression tests were conducted to examine the predictions.

ELIGIBILITY:
Inclusion Criteria:

* average score of 65 or higher in one of the BRIEF questionnaire indexes
* 70 or more in the Wechsler intelligence scale for children

Exclusion Criteria:

* psychiatric or emotional disorders, autistic disorders, physical disabilities, or neurological diseases

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Change measures from baseline, 8 weeks and 20 weeks
  an individualized outcome measure of daily activities. Each participant identified and prioritized three meaningful daily activities in which he or she perceived performance problems to be most salient. Subsequently, the participant rated each activity on a 10-point scale (1 = not able to do at all; 10 = able to do extremely well) for self-perceived performance capacity (COPM-P) and for performance satisfaction (COPM-S). Significant improvement was considered as a change of at least two points between measures.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function (BRIEF) | Change measures from baseline, 8 weeks and 20 weeks
  a parents' report consisting of 86 items, designed to evaluate the control levels of EF. Parents rate
  their child's behavior on a three-point Likert scale (1) never, (2) sometimes, (3) often. Eight scales are obtained in two indexes: a Metacognition Index (MI) containing five sub-scales; Initiate, Working Memory, Plan/Organize, Organization of Materials, Monitor; a Behavioral Regulation Index (BRI) containing three subscales: Inhibit, Shift, and Emotional Control. T-scores at or above 65 are considered clinically significant in terms of dysexecutive functions.
Behavior Rating Inventory of Executive Function (BRIEF-SR) | Change measures from baseline, 8 weeks and 20 weeks
  A self-report questionnaire used to assess EF in 11-18-year-olds. Eighty statements are included in the Behavioral Regular Index (BRI) in 4 subdomains (inhibition, shifting, emotional control and monitoring), and in 4 subdomains of the Metacognition Index (MI), (working memory, planning/organization, organization of materials, and task-complete). The BRI and MI scores are combined to constitute an overall Global Executive Composite (GEC).
  A standard score of 65 and above indicates a deficit.
Participation Measure and Environment for Children and Youth (PEM-CY) questionnaire | Change measures from baseline and 8 weeks
  questionnaire that includes 25 items focused on participation in broad types of activities at home (10 items), school (5 items), and community (10 items) setting. For each item, the parents reports on three dimensions of the child's participation: 1) frequency (8 point scale, from never (0) to daily (7); 2) level of involvement (5 point scale, from minimally involved (1) to very involved (5)); and 3) the parent's desire for change in the child's participation (yes or no, if yes, the parents can select whether he or she desire a change in frequency, level of involvement' and/or broader variety).
Computerized Penmanship Evaluation Tool (ComPET, previously referred to as POET) | Change measures from baseline and 8 weeks
  This standardized and validated non-language dependent handwriting assessment utilizes a digitizing tablet, on-line data collection and analysis software. In the current study, the adolescents were requested to copy a paragraph from a document placed in front of them onto an A4-sized lined paper affixed to the surface of a WACOM Intuos II x-y digitizing tablet (404 X 306 X 10 mm), while using a wireless electronic pen with a pressure-sensitive tip (Model GP-110). Displacement, pressure, and pen tip angle were sampled at 100 Hz via a 1300 MHz Pentium (R) M laptop computer. The primary outcome measures consisted of temporal, spatial, and pressure measures for each writing stroke, as well as performance over the entire paragraph. The task was performed in Hebrew, which progresses from right to left.
WebNeuro | Change measures from baseline and 8 weeks
  WebNeuro is a computerized neuropsychological test. It is a screening tool designed to emphasize cognitive function and its effects in different populations. This computerized assessment allows us to build a person's profile over time as there are several versions that allow for repeated measurement at several time points throughout the intervention. WebNeuro taps the following domains of cognitive function: sensorimotor, memory, executive, attention, and emotion perception (social cognition). For most tests, scoring of responses was conducted using an automated software program.
the children's cooking task (CCT) | Change measures from baseline and 8 weeks
  a performance-based evaluation developed by Chevignard et al. (2009) to assess EF and multitasking abilities. The manual, developed in French, was translated into English (Poncet et al., 2015), including the psychometric properties that were examined in two papers (Chevignard et al., 2009, 2010). Each subject was asked to prepare two simple recipes (a chocolate cake and a fruit cocktail). Ingredients and utensils were laid out on the table with an instruction page and a folder with six recipes presented in the same manner (i.e., title, illustrated list of ingredients, and numbered, illustrated preparation steps). The participants were expected to find the two correct recipes among the four distracters.
  The examiner wrote down the participant's actions and comments and then rated and classified them.